CLINICAL TRIAL: NCT05967338
Title: Comparison of Epiglottis Lifting Methods Using a McGrath Video Laryngoscope: Direct vs. Indirect
Brief Title: Glottis Visualization in Different Lifting Methods
Status: Completed | Type: Observational
Sponsor: Zonguldak Bulent Ecevit University (Other)
Responsible Party: Principal Investigator, Keziban Bollucuoglu, Principal Investigator, Zonguldak Bulent Ecevit University
Other Study IDs: 2022/12-10
Record Dates: First submitted 2023-06-01; First posted 2023-08-01 (Actual); Last update posted 2023-08-01 (Actual); Status verified 2023-07

CONDITIONS: Intubation; Glottis Visualization
Keywords: Endotrakeal intubation; Epiglottis; Glottis; McGrath MAC video laryngoscope

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Group Direct: glottis visualization in direct lifting
  Interventions: Device: using McGrath Video Laryngoscope
- Group Indirect: glottis visualization in indirect lifting
  Interventions: Device: using McGrath Video Laryngoscope

INTERVENTIONS:
Device: using McGrath Video Laryngoscope — glottis visualization in indirect and direct lifting methods by using McGrath Video Laryngoscope

SUMMARY:
Among the various types of video laryngoscopes, the McGrath MAC video laryngoscopy (VL) has become popular because it is lightweight and can be quickly and hygienically prepared by changing the blade. The aim of this study was to compare the efficacy of two different methods (direct and indirect) for epiglottis removal during visualization of the glottis using the McGrath MAC VL.

ELIGIBILITY:
Inclusion Criteria:

* ASA I-II
* general anesthesia in elective surgeries
* 18-65 years old
* body mass index (25-30)
* no risk of difficult intubation

Exclusion Criteria:

* Allergic to study drugs
* pregnant women
* emergency cases
* those with a history of difficult intubation
* those without consent
* those at risk of aspiration

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: ASA I-II, 18-65 years old patients undergoing elective surgery
Sampling Method: Probability Sample
Enrollment: 1 (Actual)
Dates: Start 2022-07-01 (Actual); Primary Completion 2023-01-30 (Actual); Study Completion 2023-03-01 (Actual)

PRIMARY OUTCOMES:
POGO scores | 1 day (through intubation )
  percentage of glottic opening

SECONDARY OUTCOMES:
Cormack-Lehane classification | 1 day (through intubation )
  assessment of laryngeal view during laryngoscopy

CONTACTS AND LOCATIONS:
Locations (1):
- Zonguldak Bülent Ecevit University, Zonguldak, Kozlu, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No